CLINICAL TRIAL: NCT01489982
Title: Treatments for Insomnia in Patients With Parkinson's Disease: A Pilot Study
Brief Title: Treatments for Insomnia in Patients With Parkinson's Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Ron Postuma, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INS-09-10
Record Dates: First submitted 2011-07-19; First posted 2011-12-12 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Parkinson's Disease; Insomnia
Keywords: Parkinson's disease; insomnia
MeSH Terms: conditions — Parkinson Disease; Sleep Initiation and Maintenance Disorders | interventions — Doxepin; zopiclone

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Light therapy (Experimental): For patients who have sleep maintenance insomnia light therapy will be administered daily. If patients suffer only from sleep onset insomnia, this light therapy will be given upon awakening in the morning. Light boxes will be provided by Litebook company. In the active therapy group, the intensity of the light will be set at 10,000 lux with a head-to-light distance of 20cm. Patients will be instructed to let the light shine indirectly on their eyes (i.e. they do not look directly at the light). Patients can be reading, eating, watching TV, etc., during the time of light therapy.
  Interventions: Device: Light box (Litebook company)
- CBT and sleep hygiene training (Experimental): This will involve education about sleep in general, giving techniques related to sleep and relaxation, tips on stress management, etc.. This will take place at the Lady Davis Institute of the Jewish General Hospital. There will be 6 weekly sessions totalling 90 minutes - most of the time this will be in a group setting, with a maximum of 6 patients per group. Light therapy will also be part of this treatment strategy. There will be separate gropus for English and French-speaking patients
  Interventions: Behavioral: CBT and sleep hygiene
- Insomnia medications (Experimental): Pharmacologic treatment will be individualized depending on patient characteristics and initial response. It will consist of two potential treatments - Doxepin or Zopiclone. Both of these agents are currently used commonly in the general population and also in PD patients. The agents will be prescribed exactly as any other medical prescription (i.e. patients will fill their own prescriptions at their own pharmacy).The decision for which agent to use will be as follows: a)If patients suffer from sleep onset insomnia (with or without sleep maintenance insomnia), or if doxepin is contraindicated, Zopiclone will be prescribedb) or b)If patients suffer from sleep maintenance insomnia only (or if Zopiclone is contraindicated), Doxepin will be the first choice agent.
  Interventions: Drug: Doxepin and Zopiclone
- Placebo intervention of light therapy (Placebo Comparator): The inactive/placebo intervention will be 30 minutes of light therapy, using red light below the threshold required to entrain light cycles. This therefore functions as a placebo condition for the active light therapy protocol. Patients be informed that some forms of light therapy will be expected to be less active, but we will not disclose what type of condition is inactive.
  Interventions: Device: Light box ( Litebook company)

INTERVENTIONS:
Device: Light box (Litebook company) — Light therapy will be administered daily for a duration of 30 minutes, starting two hours (+/- 1 hour) prior to usual bedtime
  Arms: Light therapy
Behavioral: CBT and sleep hygiene — 6 weekly sessions totalling 90 minutes
  Arms: CBT and sleep hygiene training
Drug: Doxepin and Zopiclone — Zopiclone 3.75 mg at h.s., increasing to 7.5 mg after one week if insufficient clinical effects ( and no troublesome side effects) or Doxepin 5 mg at h.s. followed by increase up to 10 mg after the first week if insufficient clinical effect (and no troublesome side effects)
  Arms: Insomnia medications
Device: Light box ( Litebook company) — The intervention will be 30 minutes of light therapy, using red light below the threshold required to entrain light cycles
  Arms: Placebo intervention of light therapy

SUMMARY:
More than half of patients with Parkinson's have troubles with insomnia. There are several treatment options for insomnia that have been studied in the general population - however, the investigators don't know if these treatments work for patients with Parkinson's. It is possible that people with Parkinson's may have different treatment responses.

The goal of this project is to test in a pilot study the tolerability and effectiveness of pharmacologic and non-pharmacologic treatments to improve insomnia in patients with Parkinson's disease. Each participant in this study will be wearing a wrist actigrapch and fill out the sleep diary. Three main treatment strategies will be tested: Placebo Light therapy, Cognitive behavioural therapy and active light therapy, and insomnia medications. The treatment that each person will receive first will be chosen randomly. If the first therapy has not been effective, participant may choose to re-enrol in the trial with one of the remaining two therapies.

DETAILED DESCRIPTION:
There are now a variety of treatments that can help to manage insomnia, including non-pharmacological and pharmacologic measures. Although many of these strategies have been proven to be effective in the general population very few studies have been conducted with Parkinson's Disease (PD) patients. Insomnia in PD has unique characteristics and pathophysiology; therefore, measures to treat insomnia in the general population may be ineffective in PD.

The goal of this project is to test in a pilot study the tolerability and effectiveness of pharmacologic and non-pharmacologic treatments to improve insomnia in patients with Parkinson's disease.

Participants will come for four visits: for screening, then in 1 week, 3 weeks and 7 weeks. Study visits should take approximately 1.5 to 2 hours. During the entire period of the study, the participant will be wearing a wrist actigraph - this is a motion sensing device the size of a wristwatch. Specific instructions how to use this device and how to use the sleep diary will explained at the first visit. Participant will also be filling out sleep diaries every day, to keep track of how many hours you sleep, etc. During each of the study visits there will be an in-depth interview, and researcher will review with the participants their sleep diaries and troubleshoot any problems.

In this trial the investigators will be testing three main treatment strategies. The treatment that the patient will receive first will be chosen randomly - this is essential to properly test our strategies. Participant will know which group he/she has been assigned to. If the first therapy has not been effective for the patient, he/she may choose to re-enroll in the trial, in which case participant will receive one of the remaining two therapies. The therapies are:

1. Light therapy, which patient will use for 30 minutes, starting at two hours (+/- 1 hour) before your usual bedtime. Light boxes will be provided by our team. Patient will be instructed how to use this light.
2. Cognitive behavioural therapy and sleep hygiene training - This will involve education about sleep in general, giving techniques related to sleep and relaxation, tips on stress management, etc.. This will take place at the Lady Davis Institute of the Jewish General Hospital. There will be 6 weekly sessions totaling 90 minutes - most of the time this will be in a group setting, with a maximum of 6 patients per group. Light therapy will also be part of this treatment strategy.
3. Insomnia medications - In this portion patient will receive medications to help them sleep. Depending on the type of patient's sleep problem, this will either be a medication called desipramine (also called Doxepin), or zopiclone (also called Imovane). Both of these medications are currently used for insomnia in people without Parkinson's. These medications will be prescribed exactly as any other medical prescription, and participant will take them as any other medical prescription.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be recruited from the Movement Disorder Clinics at the McGill University Health Center.
* Patients will be eligible for inclusion if they have a diagnosis of idiopathic PD and suffer from insomnia, defined as an SCOPA-sleep nocturnal subscore of >7.
* The insomnia must have been persistent for at least 6 months (by patient self-report).
* The subjects must speak either English or French sufficiently to fill out questionnaires.

Exclusion Criteria:

1. Use of sedative medications at night (including sedating antidepressants). Patients may be taking non-sedating antidepressants if dose is stable for 1 month.
2. Untreated restless legs syndrome, night shift work, occupational causes of abnormal sleep pattern, or other reversible causes of insomnia detected upon baseline clinical interview. If treatment of a potentially-reversible cause is unsuccessful and insomnia is persistent >3 months following treatment initiation, patients can be enrolled.
3. Insomnia is not secondary to suboptimal dopaminergic therapy. If changes to dopaminergic therapy are required after clinical interview, patients can still be eligible for inclusion if insomnia is persistent >3 months.
4. Pre-menopausal women who are not using effective methods of birth control (note that only a small minority of women with PD are pre-menopausal, so the effects of this exclusion criterion in creating gender imbalance should be minimal).
5. Dementia, defined according to PD dementia criteria as MMSE <26/30 and ADL impairment secondary to cognitive loss, or inability to understand consent process.
6. Change to dopaminergic therapy over the preceding three months.
7. Patients with very severe PD, defined as Hoehn and Yahr of 5 (i.e. nonambulatory). Provision of sleep hygiene measures, etiology of insomnia, and potential confounds in interpretation of actigraphy in immobile patients is problematic in very advanced stages of PD.
8. Insomnia is related to untreated moderate-severe depression or anxiety. Beck depression score > 20i.e, moderate depression).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
SCOPA sleep scale | 6 weeks
  The SCOPA sleep scale is a disease-specific measure that has been designed to assess sleep in PD. It is divided into two sections which address occurrence of nighttime sleep problems and daytime sleepiness in PD over the past month. It has been recommended as a scale of choice for evaluation of insomnia by the Movement Disorders Task Force for Sleep assessment in PD. A nocturnal subscale score of >7 was proposed as a cutoff to define poor sleep, based upon the global sleep assessment, a cutoff confirmed in a subsequent study.
Actigraphy | 6 weeks
  Actigraphs are motion sensing devices the size of a wristwatch, which are constantly worn by the patient. Absence of physical activity for a prolonged interval is interpreted as onset of sleep The actigraph used will be the ActiWatch Spectrum (Philips Respironics). The primary outcomes of interest with actigraphy will be total sleep time, sleep efficiency, wake after sleep onset, sleep fragmentation, and duration and number of naps (sleep onset latency will also be assessed, but will be supplemented mainly with diary, since onset latency is not reliably assessed with actigraphy).

SECONDARY OUTCOMES:
Daily sleep dairy | 6 weeks
  Daily sleep dairy is a standard assessment procedure in insomnia treatment research to collect descriptive sleep data. It is a very practical and cost-effective method for assessing insomnia when repeated measurements are needed. The following items are normally included in sleep diaries: bedtime, arising time, sleep latency, number and duration of awakenings, sleep duration, naps, medication intake, and others.
Insomnia severity Index (ISI) | 6 weeks
  This brief self-report instrument measures the patient's perception of his insomnia. It has been selected as one of the non PD-specific measures used for insomnia. The questionnaire includes 7 items that evaluate the severity of sleep initiation, the sleep maintenance, and other aspects related to insomnia. This instrument has been extensively validated in the general population.
Pittsburgh Sleep Quality Index (PSQI) | 6 weeks
  This self-rated extensively-validated questionnaire contains 19 items that are divided into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. It also tracks use of sleep medications. It is perhaps the most commonly used non-disease-specific measure of sleep quality.
Parkinson's Disease Sleep Scale (PDSS) | 6 weeks
  This questionnaire is a visual analogue scale assessing 15 features of sleep disturbance in patients with PD. It addresses overall quality of sleep, sleep onset and maintenance insomnia, nocturnal restlessness, nocturnal psychosis, nocturia, nocturnal motor symptoms, sleep refreshment, and daytime dozing. This questionnaire has been validated with PD patients. The PDSS is useful to asses overall nocturnal sleep quality in patients with PD. Its inclusion of items such as nocturnal motor symptoms and nocturia also allows it to assess potential reversible causes of insomnia.
Clinical global impression of change | 6 weeks
  Completed by both the examiner and the patient, the scale is a single question about insomnia severity that is scored as very much improved (6), much improved (5), minimally improved (4), no change (3), minimally worse (2), much worse (1), or very much worse (0).
The Krupp Fatigue Severity Scale | 6 weeks
  The fatigue severity scale measures impact of fatigue with a 9-item questionnaire, with a 7-point Likert scale for each question. It has been validated, and has been used in PD studies, including trials of excessive daytime somnolence.
Beck depression index | 6 weeks
  The Beck Depression Inventory is a self-administered scale of 21 items (scored 0-3) which assesses depression symptoms. The Beck Inventory is one of the most commonly-used scales for depression in PD, and a recent consensus panel of the Movement Disorders Society concluded it was a scale of first choice for assessing depression in PD.
Adherence to treatment | 6 weeks
  The compliance will be assessed by numerous measures. Compliance with medical therapy will be conducted by pill counts, to compare numbers of pills prescribed and taken. Compliance with sleep hygiene measures will be assessed by sleep diary and actigraphy. Compliance with light therapy will be assessed using actigraphy, which contains a light sensor.
Severity of motor manifestations (UPDRS) | 6 weeks
  This is the standard scale used for grading severity of PD. It consists of a systematic history assessing problems with motor function, cognition, psychiatric state, and side effects of medications, as well as examination rating features of PD. The UPDRS Part III examination component will be performed in the medication 'on' state at each clinical visit UPDRS Part IV will be recorded and coded separately for fluctuations and dyskinesia. Total 'off' time (in hours) will be also recorded, as assessed by clinical interview.
Quality of life (PDQ-39) | 6 weeks
  The Parkinson's Disease Questionnaire is a quality of life index for PD. It consists of a 39-item questionnaire that asks about the impact of PD on a person's motor function, gait, mood, cognition, and activities of daily living.
Adverse events | 6 weeks
  Adverse events will be queried by means of a semi structured interview - "Have you had any side effects?". The open-ended - question to researcher will be asked - "Do you think this related? Is it a serious adverse event?" That will be scored as mild =1, moderate =2 or severe=3.
Sleep Hygiene Index | 6 weeks
  This self-administered instrument contains 13 items related to diagnostic criteria for inadequate sleep hygiene according to the International Classification of Sleep Disorders. This instrument is primarily used to determine the causes of insomnia - high scores indicate more maladaptive sleep hygiene practices. The Sleep Hygiene Index has been validated in the general population and has been found to be a reliable instrument.
Dysfunctional Beliefs and Attitudes about Sleep, a brief version ( DBAS 16) | 6 weeks
  This is 16 -item self-reported questionnaire designed to evaluate various sleep/insomnia-related cognitions. These domains include expectations about sleep requirements, attributions of the causes and appraisals of the consequences of insomnia, and issues of worry and helplessness about insomnia. The DBAS -16 has been validated and has been found to be a reliable scale.
Epworth Sleepiness Scale (ESS) | 6 weeks
  This is a scale for measurement of the level of daytime sleepiness. The short questionnaire asks the subject to rate his or her probability of falling asleep on a scale of increasing probability from 0 to 3 for eight different situations.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Postuma, MD, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada